CLINICAL TRIAL: NCT02102022
Title: Phase 1/2 Study of ADI-PEG 20 Plus FOLFOX in Subjects With Advanced Gastrointestinal Malignancies Focusing on Hepatocellular Carcinoma
Brief Title: Ph 1-2 Study ADI-PEG 20 Plus FOLFOX in Subjects With Advanced GI Malignancies Focusing on Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLARIS2013-001
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2019-05

CONDITIONS: Advanced Gastrointestinal (GI) Malignancies; Hepatocellular Carcinoma; Gastric Cancer; Colorectal Cancer
Keywords: argininosuccinate synthetase; arginine; arginine deiminase
MeSH Terms: conditions — Neoplasms; Carcinoma, Hepatocellular; Stomach Neoplasms; Colorectal Neoplasms | interventions — ADI PEG20

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- ADI-PEG 20 plus modified FOLFOX6 (Experimental): Dose: 36 mg/m2 given weekly
  Route of Administration: Intramuscular (IM)
  In combination with modified FOLFOX6, every 2 weeks, intravenous (IV) / IV bolus
  Interventions: Drug: ADI-PEG 20 plus modified FOLFOX6

INTERVENTIONS:
Drug: ADI-PEG 20 plus modified FOLFOX6
  Other Names: pegargiminase

SUMMARY:
Phase 1: Assessment of safety and tolerability of ADI-PEG 20 in combination with folinic acid (leucovorin), fluorouracil and oxaliplatin (FOLFOX) in advanced GI malignancies.

Phase 2: Assessment of the objective response rate (ORR), measured by RECIST 1.1 criteria as assessed by blinded independent central review (BICR).

DETAILED DESCRIPTION:
Phase 1:The primary objective of the dose escalation portion of this study was to assess the safety and tolerability of ADI-PEG 20 in combination with folinic acid (leucovorin), fluorouracil (5-FU), and oxaliplatin (mFOLFOX6) in advanced GI malignancies. The primary objective of the maximum tolerated dose (MTD) expansion phase (recommended phase 2 dose [RP2D]) of this study was to determine preliminary estimates of efficacy, measured by RECIST 1.1 criteria, for ADI-PEG 20 in combination with FOLFOX in hepatocellular carcinoma (HCC), gastro-esophageal cancer (GEC), and colorectal cancer (CRC).

Phase 2: The primary objective of this single arm trial is ORR. Based on a two-sided exact test of a one-sample proportion with an alpha of 0.05, under a presumed ORR of 22%, there is 80% power to yield 95% confidence interval of 15-26%, which will require 46 objective responses in 225 subjects. A futility analysis will be described in the Statistical Analysis Plan.

ELIGIBILITY:
Phase 2 HCC Subjects:

Inclusion Criteria:

1. Advanced histologically or cytologically proven HCC (except with prior liver transplantation).
2. Treatment with at least 2 prior systemic therapy regimens.
3. Child-Pugh grade A. Child-Pugh status should be determined based on clinical findings and laboratory data during the screening period (Appendix C).
4. Measurable disease using RECIST 1.1 criteria (Appendix A). At least 1 measurable lesion must be present. Subjects who have received local-regional therapies are eligible, provided that they have either a target lesion which has not been treated with local therapy and/or the target lesion(s) within the field of the local regional therapy has shown an increase of ≥ 20% in size. Local-regional therapy must be completed at least 4 weeks prior to the baseline CT scan.
5. ECOG performance status of 0 - 1.
6. Expected survival of at least 3 months.
7. Age ≥ 18 years.
8. Fully recovered from any prior surgery and no major surgery within 4 weeks of initiating treatment. Surgery or procedure for placement of vascular access devices is exempt from this period.
9. Subjects must agree to use at least one form of highly effective contraception or agree to refrain from intercourse for the duration of the study. Contraceptive use must be continued until at least 30 days after the last administration of ADI-PEG 20 and at least 90 days after the last administration of FOLFOX. For female subjects, a serum human chorionic gonadotropin (HCG) pregnancy test must be negative before entry into the study. If HCG pregnancy test is positive, further evaluation to rule out pregnancy must be performed according to GCP before this patient is claimed eligible.
10. Informed consent must be obtained prior to study initiation.
11. No concurrent investigational studies are allowed.
12. Total bilirubin < 1.5 x upper limit of normal range.
13. Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x upper limit of normal range.
14. Absolute neutrophil count (ANC) > 1500/μL.
15. Platelets > 75,000/μL.
16. Serum uric acid ≤ 8 mg/dL (with or without medication control).
17. Serum creatinine ≤ 1.5 x the upper limit of normal range, or, if serum creatinine >1.5 x the upper limit of normal range, then the creatinine clearance must be ≥ 60 mL/min/1.73 m2 (calculated using the Jelliffe equation: calculated creatinine clearance = 98 - 0.8 [age (yrs.) - 20] /serum creatinine (x 0.9 if female).
18. Brain metastases are allowed if well controlled and without seizures.
19. Serum albumin level ≥ 2.8 g/dL.
20. Prothrombin time (PT)-international normalized ratio (INR): PT <6 seconds above control or INR <1.7. Subjects on Coumadin anti-coagulants are to receive only 1 point for their INR status.
21. Subjects with active hepatitis B or C on anti-viremic compounds may remain on such treatment, except for interferon.

Exclusion Criteria:

A subject will not be eligible for study participation if he/she meets any of the exclusion criteria:

1. Serious infection requiring treatment with systemically administered antibiotics at the time of study entrance, or an infection requiring systemic antibiotic therapy within 7 days prior to the first dose of study treatment.
2. Pregnancy or lactation.
3. Expected non-compliance.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV), cardiac arrhythmia, or psychiatric illness.
5. Subjects who have had any anticancer treatment prior to entering the study and have not recovered to baseline (except alopecia) or ≤ Grade 1 AEs, or deemed irreversible from the effects of prior cancer therapy. AEs > Grade 1 that are not considered a safety risk by the Sponsor and investigator may be allowed upon agreement with both.
6. Subjects with history of another primary cancer, including co-existent second malignancy, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor with no known active disease present or in the opinion of the investigator will not affect patient outcome.
7. Subjects who had been treated with ADI-PEG 20 previously.
8. History of seizure disorder not related to underlying cancer.
9. Known HIV positivity (testing not required).
10. Known allergy to pegylated compounds.
11. Known allergy to E. coli drug products (such as GMCSF).
12. Known allergy to oxaliplatin or other platinum compounds.
13. Prior grade 2 or higher neuropathy from prior platinum unless neuropathy is currently ≤ grade 1.
14. Contraindications to fluorouracil

    1. Subjects with poor nutritional state.
    2. Known depressed bone marrow function.
    3. Subjects with potentially serious infections.
    4. Known allergy to fluorouracil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-11; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Date of first study drug administration to the date of disease progression (measured every 8 weeks) or death (whichever occurs first), up to 24 months
  The percent of subjects who exhibit each level of tumor response, measured by RECIST 1.1 criteria as assessed by blinded independent central review.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Date of first study drug administration to the date of disease progression (measured every 8 weeks) or death (whichever occurs first), 12 months anticipated
  Time from the first dose until objective tumor progression or death from any cause
Overall survival (OS) | Date of first study drug administration through study completion
  The time from first treatment with ADI-PEG 20 until death or censoring
Duration of response (DoR) | From date of first response until the date of documented progression or date of death, 12 month in average
  the time in weeks between the first occurrence of objective response and the development of progressive disease or death
Disease control rate (DCR) | Date of first study drug administration to the date of disease progression (measured every 8 weeks) or death (whichever occurs first), up to 24 months.
  the proportion of subjects at each post-baseline assessment who exhibit tumor response of complete response, partial response or stable disease
Pharmacodynamics | At week 1, 5, 9, 13, 17, 21 prior to ADI-PEG 20 administration
  Blood levels of arginine and citrulline
Pharmacokinetics Variable | At week 1, 5, 9, 13, 17, 21 prior to ADI-PEG 20 administration
  Peripheral blood levels of ADI-PEG 20
Immunogenicity | At week 1, 5, 9, 13, 17, 21 prior to ADI-PEG 20 administration
  antibodies to ADI-PEG 20
AFP (alpha feto-protein) changes | At baseline, week3, 7, 11, 15, 19, 23 and end of treatment
  Maximal percent changes of AFP during the course of study compared to AFP at baseline

CONTACTS AND LOCATIONS:
Overall Officials: James Harding, MD, Principal Investigator — Memorial Sloan-Kettering Cancer Center (MSKCC)
Locations (35):
- United States (10):
  - California Pacific Medical Center, San Francisco, California
  - Emory University, Atlanta, Georgia
  - The University of Chicago Medical Center, Chicago, Illinois
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Washington, Seattle, Washington
- China (2):
  - The Chinese People's Liberation Army 81 Hospital, Nanjing, Jiangsu
  - West China Hospital, Sichuan University, Chengdu, Sichuan
- Italy (2):
  - IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - National Cancer Institute of Napoli IRCCS G. Pascale, Napoli
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Pusan National University Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
- Taiwan (11):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation - Kaohsiung, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - Chi Mei Hospital, Liouying, Tainan
  - Mackay Memorial Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
- United Kingdom (4):
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral
  - Royal Free Hospital, London
  - Guy's & St Thomas' NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester